CLINICAL TRIAL: NCT03592810
Title: Multi-center Observational Study to Assess Optimal ECMO Settings During the First Hours of Extracorporeal Cardiopulmonary Resuscitation
Brief Title: Observational Study to Assess Optimal ECPR Settings After Resuscitation
Acronym: MOFE
Status: Completed | Type: Observational
Sponsor: Erasmus Medical Center (Other)
Responsible Party: Principal Investigator, Loes Mandigers, MD, Principal Investigator, Erasmus Medical Center
Other Study IDs: NL60632.078.17
Record Dates: First submitted 2018-06-19; First posted 2018-07-19 (Actual); Last update posted 2021-02-23 (Actual); Status verified 2021-02

CONDITIONS: Extracorporeal Cardiopulmonary Resuscitation; Cardiac Arrest
MeSH Terms: conditions — Heart Arrest

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- ECPR: All patients who received ECMO placement during cardiopulmonary resuscitation (ECPR)
  Interventions: Other: Settings of the extracorporeal membrane oxygenation (ECMO)

INTERVENTIONS:
Other: Settings of the extracorporeal membrane oxygenation (ECMO) — Compare the settings of the ECMO in different European hospitals and relate them to cerebral saturation and neurological outcome, using Cerebral Performance Category (CPC) score
  Other Names: Measurements of cerebral saturation

SUMMARY:
Rationale: Veno-arterial extracorporeal membrane oxygenation (vaECMO) during cardiopulmonary resuscitation (ECPR) might improve outcome after cardiac arrest. However, it is well established that reperfusion injury of the brain can cause microvascular and endothelial dysfunction, leading to cellular necrosis and apoptosis. While performing ECPR, following the European resuscitation guidelines, it is yet unknown how to set the ECMO settings in order to minimize ischemia-reperfusion injury of the brain.

Objective: In this study, we want to elaborate on the optimal ECMO settings in the first three hours after initiation of ECPR.

Study design: Prospective, multi-centre, observational study Study population: All patients receiving ECPR in the age between 18 and 70 years, with low flow duration<60min and receiving cerebral oximetry monitoring Intervention: application of an adhesive regional oximetry sensor on the patient's forehead and withdrawal of 12 ml extra blood in all patients.

Main study parameters/endpoints: Cerebral Performance Category at 6 months. Neuron-specific enolase (NSE) will be determined from routine blood drawings.

ELIGIBILITY:
Inclusion Criteria:

* Witnessed cardiac arrest or signs of life during CPR (such as gasping or movement)
* Age>18 and < 70 years
* Duration of low-flow < 60 min before decision to proceed with ECPR
* High quality CPR (defined as end-tidal carbon dioxide (CO2et) >10 mmHg) provided for a minimum of 15 minutes without return of spontaneous circulation (ROSC)
* Presumed cardiac cause of cardiac arrest (such as Chest pain before collapse, ventricular tachycardia/ventricular fibrillation (VT/VF) as initial rhythm or ST-elevation on ECG)
* Cerebral oxymetry monitoring initiated during CPR preceding ECPR

Exclusion Criteria:

* Patients with a GCS<15 before CPR.
* Known pre-arrest cerebral performance category CPC ≥ 3
* Presumed noncardiac cause
* Unwitnessed collapse
* Suspected or confirmed pregnancy
* ROSC within 5 minutes of Advanced cardiopulmonary life support (ACLS) performed by emergency medical service (EMS) team
* Conscious patient
* Known bleeding diathesis or suspected or confirmed acute or recent intracranial bleeding
* Suspected or confirmed acute stroke
* Known severe chronic organ dysfunction or other limitations to therapy
* "Do not resuscitate" order or other circumstances that make 180 day survival unlikely

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adult patients receiving ECPR will be included. The decision to perform an ECPR is made by the local protocol and clinical judgment of the attending physician.
Sampling Method: Non-Probability Sample
Enrollment: 26 (Actual)
Dates: Start 2018-07-18 (Actual); Primary Completion 2020-03-01 (Actual); Study Completion 2020-09-30 (Actual)

PRIMARY OUTCOMES:
CPC score 6 months | 6 months
  To prospectively identify parameters correlated with Cerebral Performance Category (CPC)* ≤ 2

SECONDARY OUTCOMES:
CPC score discharge | 6 months
  Parameters correlated with a CPC* ≤ 2
Glasgow coma scale (GCS) day 28 | 6 months
  Parameters correlated with a GCS>13
GCS total | 6 months
  Parameters correlated with a GCS > 13
28 day mortality | 6 months
  Parameters correlated to 28 days mortality
Hospital survival | 6 months
  Parameters correlated to hospital survival

CONTACTS AND LOCATIONS:
Overall Officials: Dinis dos Reis Miranda, PhD, MD, Principal Investigator — Erasmus Medical Center
Locations (1):
- ErasmusMC, Rotterdam, Netherlands

IPD SHARING:
Plan to Share IPD: No